CLINICAL TRIAL: NCT07217288
Title: Effectiveness of Complete Decongestive-versus Non-pneumattic- Compression Therapy in Patients With Post-mastectomy Lymphedema
Brief Title: Complete Decongestive Therapy Versus Non-pneumatic Compression Therapy in Post Mastectomy Lymphedema
Acronym: CDT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Collaborators: University of Lahore (Other)
Responsible Party: Principal Investigator, Sahar Fatima, Sahar Fatima, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/12/0042; U1111-1329-7030 (Registry Identifier: World Health Organization)
Record Dates: First submitted 2025-10-09; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Lymphedema, Breast Cancer; Mastectomy Related Lymphedema; Post Mastectomy Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Complete Decongestive Therapy (CDT) and Routine Physical Therapy (Active Comparator): Group A: Complete Decongestive Therapy (CDT) and Routine Physical Therapy:
  Manual Lymphatic Drainage (MLD)
  * Duration: 30 minutes/session
  * Frequency: 5 days/week
  * Technique: Performed by a certified lymphedema therapist
  * Areas: Neck, axilla, trunk, and affected limb
  * Total treatment time: 8 weeks 2. Compression Bandaging
  * Type: Multi-layer short-stretch bandaging
  * Application: After MLD in each session
  * Worn Duration: 22-23 hours/day
  * Reapplied Daily: Yes 3. Skin Care
  * Duration: 10 minutes/session
  * Components:
    * Inspection of skin
    * Use of pH-neutral moisturizers
    * Infection prevention education 4. Exercise Therapy (Routine Physiotherapy)
  * Type: Gentle, active ROM and resistance exercises (e.g., shoulder mobility, grip strengthening)
  * Duration: 20 minutes/session
  * Progression: Gradually increase intensity over 8 weeks
  Interventions: Other: Complete Decongestive therapy
- Group B: Non-pneumatic compression device (NPCD) and Routine Physiotherapy (RPT) (Experimental): Subjects will be taught how to apply the device themselves, including placement, duration of use, and turning it on/off. All subjects will be instructed to wear the device for up to 40 minutes per day and to continue their usual activity during use. Routine Physical Therapy:
  * Type: Gentle, active ROM and resistance exercises (e.g., shoulder mobility, grip strengthening)
  * Duration: 20 minutes/session
  * Progression: Gradually increase intensity over 8 weeks
  Interventions: Device: Non Pneumatic compression device

INTERVENTIONS:
Device: Non Pneumatic compression device — Non-Pneumatic Compression Device (NPCD) is a wearable, portable system providing gradient sequential compression through shape-memory alloy actuators instead of air pressure. Frequency: 5 sessions per week for 8 weeks.
  Intensity: Moderate, rhythmic static and dynamic compression applied distally to proximally, allowing safe lymphatic drainage.
  Time: 40 minutes per session, once daily.
  Arms: Group B: Non-pneumatic compression device (NPCD) and Routine Physiotherapy (RPT)
Other: Complete Decongestive therapy — Complete Decongestive Therapy (CDT), is the gold-standard, non-invasive treatment for lymphedema. It combines manual lymphatic drainage (MLD), compression bandaging, exercise therapy, and skin care to reduce limb swelling and improve lymphatic flow.
  Frequency: 5 sessions per week for 8 weeks. Intensity: Gentle manual drainage with multilayer compression Time: 60 minutes per session. Type: Therapist-guided manual and compression therapy followed by self-management.
  CDT aims to decongest the limb, prevent fibrosis and infection, and enhance mobility and quality of life in post-mastectomy lymphedema patients.
  Arms: Complete Decongestive Therapy (CDT) and Routine Physical Therapy

SUMMARY:
The aim of the study is to compare the effectiveness of Complete Decongestive Therapy and Non-Pneumatic Compression Therapy, both combined with routine physical therapy, in reducing pain and edema volume, improving range of motion, respiratory function, inflammatory markers, and overall quality of life in patients with post-mastectomy lymphedema.

DETAILED DESCRIPTION:
Post-mastectomy lymphedema (PML) is a chronic, progressive, and disabling complication affecting breast cancer survivors due to disruption of lymphatic drainage following surgery or radiotherapy. It leads to swelling, pain, restricted range of motion, recurrent infections, and reduced quality of life.

Complete Decongestive Therapy (CDT) - a multimodal approach involving manual lymphatic drainage, compression bandaging, skin care, and exercise - is currently the gold standard for lymphedema management. However, CDT is time-consuming, therapist-dependent, and often poorly tolerated or inaccessible for long-term self-management.

Non-Pneumatic Compression Therapy (NPCD) is a newer, portable, and wearable device that provides gradient sequential compression while allowing mobility and daily activity during treatment. It potentially improves adherence, comfort, and patient satisfaction.

Limited comparative research exists evaluating the relative effectiveness of CDT and NPCD in post-mastectomy lymphedema. This study aims to fill this gap and determine which approach produces superior clinical and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Females with age between 30 to 60 years. (Monticciolo et al., 2021)
* Females with unilateral mastectomy post three months of surgery. (Shen et al., 2023) 21
* A volume difference to the circumferential measurements between the affected and unaffected upper extremities of more volume difference>10%.
* Completed chemotherapy and/or radiation therapy. (Borman, Yaman, Yasrebi, İnanlı, & Dönmez, 2022)

Exclusion Criteria:

* Systemic disorders that might contraindicate the use of sequential compression therapy i.e. chronic kidney disease with renal failure, Congestive heart failure, neurological disorders, respiratory disorders.
* Presence of active cellulitis, open and partially healed wounds.
* Patients with lipedema
* Active or recurrent cancer (defined as < 3 months since completion of cancer therapy)
* An acute infection within the previous 4 weeks
* Active venous thromboembolic edema
* Pregnant women and women who are planning or nursing at study entry.
* Patients who had participated in any clinical trial of an investigational substance or device during the previous 30 days
* Potential patients with a cognitive or physical impairment that would interfere with appropriate use of the device. (Rockson, Whitworth, et al., 2022)

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-10-26 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain measured by visual analogue scale. | Assessment will be done at baseline, 4th week and 8th week.
  Lymphedema-related symptoms (pain, pressure, heaviness and hardness). The visual analogue scale (VAS) is a validated, subjective measure for acute or chronic pain. Scores are based on self-reported measures of symptoms from 0-10 score. With zero "no pain" and 10 "worst pain". Test-rater reliability has been shown to be good, but higher among literate (r= 0.94, P=0.001) than illetrate patients (r= 0.71, P=0.001).

SECONDARY OUTCOMES:
Edema volume by water displacement method | Assessment will be done at baseline, 4th week and 8th week.
  In the volumetric assessment of lymphedema, the water displacement method involves submerging the affected limb in a water-filled container and measuring the amount of water displaced. The volume change will be determined by subtracting the initial water volume from the final volume after immersing the limb, providing an estimation of limb volume.
Quality of life measured by Lymphoedema Functioning Disability and health questionnaire for the upper limb (Lymph-ICF-UL) | Assessment will be done at baseline, 4th week and 8th week
  Quality of life will be assessed using Lymphoedema Functioning Disability and health questionnaire for the upper limb (Lymph-ICF-UL). The Lymph-ICF-UL consists of 29 questions. The questionnaire consists of 5 domains: the physical function domain contains 7 questions; the mental function domain contains 4 questions; the household domain contains 4 questions; the mobility domain contains 8 questions; and the life/ social life domain contains 6 questions. Each question has to be scored on an 11-point scale (0 to 10). The anchor points for the physical and mental function domain and household domain are 'not at all' and 'a lot'. Those for the mobility and life domain/ social life domain are 'very well' and 'not at all'. The patient has to score his/ her average problems in functioning (i.e. impairments in function and activity limitations and participation restrictions) due to the upper limb lymphoedema.
Functional mobility measured by upper extremity functional index | Assessment will be done baseline, 4th week and 8th week
  The Upper Extremity Functional Index used for measuring the functional mobility of patients with breast related lymphedema. The UEF consists of 20 items, each scored on a 5-point Likert scale ranging from: 0 = Extreme difficulty or unable to perform activity, 1 = Quite a bit of difficulty, 2 = Moderate difficulty, 3 = A little bit of difficulty, 4 = No difficulty. The total score ranges from 0 to 80, with higher scores indicating greater functional ability.
Upper limb range of motion measured by goniometer | Assessment will be done at baseline, after 4th week and 8th week
  The shoulder flexion ROM will be assessed using a 12-inch plastic goniometer. The measurement will be taken with the patient in supine lying with knees flexed, the palm facing medially, and thumbs up. The assessor stood at the side of the affected arm to perform the measurement, with the goniometer axis placed on the middle of the humeral head laterally, the stationary arm parallel with the trunk, and the moveable arm in line with the midline of the humerus. The patient will be instructed to perform flexion (with elevation) of both shoulders to avoid compensatory movement of the affected side. The angle of maximum shoulder flexion measured by the goniometer will be recorded in degrees (°). The intrarater reliability for assessing shoulder flexion ROM using a goniometer has been reported to be excellent (ICC = 0.95, 95% CI = 0.89-0.98)
Respiratory functions measured by spirometer | Assessment will be done baseline, 4th week and 8th week
  Spirometric tests will be used as an objective assessment of respiratory functions. Lung capacity and respiratory muscle strength will be assessed according to the criteria of the American Thoracic Society. During the assessment, participants will be asked to sit with their arms crossed, with clips on their noses. Assessments will be conducted with the filter with in the disposable mouth piece. Evaluation of lung capacity will be started with normal breathing, continued with deep inspirations, and ended with a strong and long expiration from the participant. For the first second, the values of forced expiration volume (FEV1) and forced vital capacity (FVC) will be recorded. The best values will be recorded after repeating the assessments three times. For maximal inspiratory pressure (MIP), the nose of the participant will first closed with a clip; after the forced expiration, maximal inspiration will be recorded.
Inflammatory markers CK, CRP, IL-6, and TNF-α | Assessment will be done at baseline, after 4th week and 8th week
  Venous blood samples will be collected from the non-affected arm by a qualified phlebotomist immediately prior to and after the end of the treatment sessions. Because of risk reduction guidelines (ie, guidelines to minimize injections to the hand and arm), researchers aimed to minimize patient burden by allowing only two blood withdrawals before and after the study. This sampling time point will allow reserachers to determine whether a robust and sustained inflammatory response will be induced by exercises. Samples will be assessed for CK, CRP, IL-6, and TNF-α using standard techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Care Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No